CLINICAL TRIAL: NCT00230737
Title: Melatonin Randomized Trial for Insomnia in the Elderly
Brief Title: Effects of Melatonin on Insomnia Symptoms in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nalaka Gooneratne (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Nalaka Gooneratne, Associate Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AT001521-01A1 (NIH); R01AT001521-01A1 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-10-03 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Aged; Sleep; Insomnia; Melatonin; Neurobehavioral Manifestations; Circadian Rhythms; Human; Polysomnography; Elderly
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neurobehavioral Manifestations | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Melatonin 0.4 mg
  Interventions: Drug: Melatonin 0.4 mg
- B (Experimental): Melatonin 4.0 mg
  Interventions: Drug: Melatonin 4.0 mg
- C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 0.4 mg
  Arms: A
Drug: Melatonin 4.0 mg
  Arms: B
Drug: Placebo
  Arms: C

SUMMARY:
This study will determine whether melatonin tablets will increase the sleep of older adults with insomnia.

DETAILED DESCRIPTION:
Melatonin is a hormone secreted predominantly during the sleep period, suspected to have a strong link to the circadian sleep-wake cycle. Melatonin is also available in a pill form and, when administered during the day, tends to have a sedative effect. Clinical trials that have examined the nocturnal effects of melatonin have focused on patients of any age who have insomnia, regardless of their endogenous melatonin levels. Data indicate, however, that individuals with low endogenous melatonin levels may be more responsive to exogenous melatonin. Generally, melatonin levels decrease with age; therefore, older individuals with insomnia represent an ideal population in which to study the effects of exogenous melatonin on sleep. This study will provide older adults with insomnia melatonin tablets to determine whether the tablets will increase their sleep.

Participation in this study will last 10 weeks and will comprise overnight visits at 2 timepoints, the beginning of Week 1 and the end of Week 6. At study entry, participants will be admitted to the General Clinical Research Center for a 3-night stay, beginning with an overnight urine screen to confirm low melatonin levels. Participants will also be asked to begin a sleep diary documenting their sleep quality and quantity; the diary will be used throughout the study. During Night 1 at the clinic, participants will have urine samples collected throughout the night. Night 2 will be an adaptation night to allow participants to get used to their surroundings. On Night 3, participants will have sensors attached to their bodies and a polysomnograph machine will be used to measure their sleep efficiency. Participants with sleep efficiencies of 80% or higher will complete their study participation. Participants with sleep efficiencies less than 80% will be randomly assigned to one of three study treatments daily for 6 weeks: high-dose melatonin (4.0 mg), low-dose melatonin (0.4 mg), or placebo. Participants will have study visits at Weeks 1, 3, and 6 to monitor for adverse events. After 6 weeks, participants will have 2 more overnight clinic visits that will be identical to Nights 2 and 3 from the beginning of the study. Sleep questionnaires, cognitive tests, and psychomotor tests will be used to assess participants at the beginning of the study, after 6 weeks, and at the end of the study. One month after the end of the study, participants will have a follow-up visit to be reassessed for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* History of insomnia
* Low melatonin levels at study entry

Exclusion Criteria:

* History of sleep apnea (temporary cessation of breathing during sleep)
* Diagnosis of restless legs syndrome
* Current alcohol or substance abuse
* Dementia
* Anemia
* Liver disease
* Leukemia or lymphoma
* Asthma

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka S. Gooneratne, MD,MSc, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Gooneratne NS, Edwards AY, Zhou C, Cuellar N, Grandner MA, Barrett JS. Melatonin pharmacokinetics following two different oral surge-sustained release doses in older adults. J Pineal Res. 2012 May;52(4):437-45. doi: 10.1111/j.1600-079X.2011.00958.x. Epub 2012 Feb 21. PMID 22348451

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Low Dose: Melatonin 0.4 mg
- B: High Dose: Melatonin 4.0 mg
- C: Control: Placebo
Period: Overall Study
Arm/Group | A: Low Dose | B: High Dose | C: Control
Started | 9 | 10 | 8
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Low Dose | B: High Dose | C: Control | Total
Number analyzed (Participants) | 9 | 10 | 8 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (5.9) | 75.7 (4.7) | 75.1 (6.2) | 74.6 (5.6)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 7 | 7 | 20
  Male | 3 | 3 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Peak Melatonin Level
Description: Pharmacokinetic analysis of maximum melatonin level
Time Frame: day 42
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | A: Low Dose | B: High Dose | C: Control
Number analyzed (Participants) | 9 | 10 | 8
pg/ml | 405 (93) | 3999 (700) | 52 (8.1)
Statistical Analysis 1: Comparison: A: Low Dose vs B: High Dose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 3594

ADVERSE EVENTS:
Arm/Group | A: Low Dose | B: High Dose | C: Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
Study did not meet total recruitment targets

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No